CLINICAL TRIAL: NCT03766074
Title: Evaluation of Vitamin D Supplementation Effects on Serum 25(OH)D3, PTH, Pro-inflammatory Biomarkers and Neurotransmitters Involved in Depression, and Depression Status in Depressive Patients
Brief Title: Vitamin D Supplementation in Patients With Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tirang R. Neyestani, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Tirang R. Neyestani, Ph.D., Tirang R. Neyestani, Ph.D. Professor, National Nutrition and Food Technology Institute
Organization: National Nutrition and Food Technology Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 784
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Depression
Keywords: vitamin D- Depression- Cholecalciferol-
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): vitamin D supplement every other week
  Interventions: Dietary Supplement: vitamin D supplement
- control (Placebo Comparator): Placebo every other week
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: vitamin D supplement — The intervention group receives 50000 IU of vitamin D every 2 weeks as vitamin D supplements for 8 weeks, provided monthly.
  Arms: Intervention
Dietary Supplement: Placebo — placebo
  Arms: control

SUMMARY:
Groups (intervention group receives 50000 IU vitamin D and control group receives placebo) through a random allocation. After 8 weeks, blood sample will be collected from each participant. The studied indices (inflammatory (IL-1β, IL-6, hs-CRP), PTH, platelet serotonin, serum oxytocin, serum 25(OH) D, depression status and anthropometry indices) will be evaluated at beginning and end of interventional period.

DETAILED DESCRIPTION:
In this double-blind randomized clinical trial, 60 patients aged 18-60y referred to Baharlou hospital with a history of mild to moderate depression diagnosed by a psychiatrist will be presented to the researcher. After receipt of a signed informed consent form, eligible patients will participate. A general demographic questionnaire will be completed by an interviewer. Individuals are randomly divided into intervention and control groups. A 10-ml venous blood sample will be collected from each participant. The intervention group receives 50000 IU of vitamin D every 2 weeks as vitamin D supplements for 8 weeks, provided monthly. The control group receives placebo. The drug schedule of both groups (if any) will be unchanged according to the prescribing physician. After 8 weeks, blood sample will be collected from each participant. The studied indices (inflammatory (IL-1β, IL-6, hs-CRP), PTH, platelet serotonin, serum oxytocin, serum 25(OH) D, depression status, anthropometry indices) will be evaluated at beginning and end of interventional period. Data will be analyzed by statistical tests.

ELIGIBILITY:
Inclusion Criteria:

* age: 18 to 60 y
* Having mild to moderate depression

Exclusion Criteria:

* Having a history of heart infarction
* Having a history of angina
* Having a history of stroke
* Having a history of kidney stones
* Having a history of high blood pressure (systolic blood pressure higher than 174 or diastolic blood pressure higher than 104 mm Hg)
* Having a history of liver disease
* Having a history of hyperparathyroidism
* Pregnancy and/or lactation
* Reproductive-aged women (under 50 years old) who are not receiving adequate contraception
* Consuming nutritional supplement containing vitamin D from 2 months ago
* Not willing to continue the study
* Failure to follow the Supplemental Program

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-06 (Actual); Primary Completion 2019-04 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
significant change (mean±SD) in vitamin D status | baseline and 8 weeks after intervention
  The serum concentration of 25(OH) D (nmol/L) will be measured at baseline and 8 weeks after intervention. normal range is 25-162 nmol/L

SECONDARY OUTCOMES:
significant change (mean±SD) in serum concentration of IL-1β and IL-6. | baseline and 8 weeks after intervention
  The serum concentration of IL-1β and IL-6 (pg/mL) will be measured at baseline and 8 weeks after intervention.
significant change (mean±SD) in serum concentration of hs-CRP | baseline and 8 weeks after intervention
  The serum concentration of hs-CRP (mg/L) will be measured at baseline and 8 weeks after intervention. normal range is 0.3-8.6 mg/L.
significant change (mean±SD) in serum concentration of bone biomarker | baseline and 8 weeks after intervention
  The serum concentration of parathormone (PTH) (pg/mL) will be measured at baseline and 8 weeks after intervention. normal range is 10-65 pg/mL.
significant change (mean±SD) in platelet serotonin concentration (ng/10^9 platelets) | baseline and 8 weeks after intervention
  The platelet serotonin concentrations (ng/10^9 platelets) will be measured at baseline and 8 weeks after intervention. normal range is 154-1086.
significant change (mean±SD) in serum concentration of oxytocin (µU/mL) | baseline and 8 weeks after intervention
  The serum concentrations of oxytocin (µU/mL) will be measured at baseline and 8 weeks after intervention. normal range is : males:1.1-1.9, females (non-pregnant): 1.0-1.8
significant change (mean±SD) in depression status | baseline and 8 weeks after intervention
  Depression status will be measured by using Beck questioner at baseline and 8 weeks after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Tirang R. Neyestani, Ph.D, Study Chair — National Nutrition and Food Technology Research Institute
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehrān, Tehran Province, Iran

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kaviani M, Nikooyeh B, Etesam F, Behnagh SJ, Kangarani HM, Arefi M, Yaghmaei P, Neyestani TR. Effects of vitamin D supplementation on depression and some selected pro-inflammatory biomarkers: a double-blind randomized clinical trial. BMC Psychiatry. 2022 Nov 11;22(1):694. doi: 10.1186/s12888-022-04305-3. PMID 36368945